CLINICAL TRIAL: NCT02022852
Title: Efficacy and Safety of Neoadjuvant Chemo-chemoradio-chemo Sequential Therapy in Locally Advanced Mid/Low Rectal Cancer: a Phase II Trial
Brief Title: Neoadjuvant Sequential Therapy in Locally Advanced Mid/Low Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Binbin Cui, Director of Abdominal Surgery Department, Harbin Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HarbinMU-BCui-001
Record Dates: First submitted 2013-12-09; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Concurrent Chemoradiotherapy; Sequential Therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concurrent chemoradiotherapy (Active Comparator): Capecitabine neoadjuvant concurrent radiochemotherapy and XELOX adjuvant therapy
  Interventions: Drug: Capecitabine
- Sequential therapy (Experimental): XELOX/capecitabine/XELOX neoadjuvant chemo-chemoradio-chemo sequential therapy and XELOX adjuvant therapy
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: Capecitabine — 50Gy, 2Gy/day per time, 5 days a week, for 5 weeks+capecitabine 850mg/m2 bid on the day accept radiotherapy. Rest for 8 weeks and surgery followed.
  Arms: Concurrent chemoradiotherapy
Drug: XELOX — XELOX 2 cycles (oxaliplatin 130mg/m2 ivgtt 2-6h day 1,capecitabine 1000 mg/m2 bid day 1-14 repeat every 3 weeks) → 50Gy, 2Gy/day per time, 5 days a week, for 5 weeks+capecitabine 850mg/m2 bid on the day accept radiotherapy → XELOX 1 cycle. Rest for 2 weeks and surgery followed.
  Arms: Sequential therapy

SUMMARY:
Compared curative effect，safety and compliance between concurrent chemoradiotherapy and chemo-chemoradio-chemo sequential therapy in locally advanced mid/low rectal cancer.

DETAILED DESCRIPTION:
The patients were divided into two arms according to the defined conditions (pathology rectal adenocarcinoma；distal distance of tumor from anal verge < 10cm；TNM staging T3-4N0-2；no distant metastasis；Karnofsky score≥70) in this prospective, single center, open, non randomized trail (arm A:concurrent chemoradiotherapy, arm B:sequential therapy). Regimens:Arm A:50Gy,2Gy/day per time, 5 days a week, for 5 weeks. +capecitabine 850mg/m2 bid on the day accept radiotherapy. Rest for 8 weeks. Arm B: XELOX 2 cycles (oxaliplatin 130mg/m2 ivgtt 2-6h day 1, capecitabine 1000 mg/m2 Bid day 1-14, repeat every 3 weeks ) → 50Gy,2Gy/day per time, 5 days a week, for 5 weeks.+capecitabine 850mg/m2 bid on the day accept radiotherapy → XELOX 1 cycle. Rest for 2 weeks. Evaluate pre chemotherapy, pre radiotherapy and pre surgery individually. Surgeries followed TME(total mesorectal excision) and PANP(pelvic autonomic nerve preservation) for patients in both arms. Take pathological evaluation of tumors. Take XELOX therapy till 6-8 cycles(pre and after surgery total). Follow up according the schedule.

ELIGIBILITY:
Inclusion Criteria:

* Pathology rectal adenocarcinoma
* Distal distance of tumor from anal verge < 10cm
* TNM staging T3-4N0-2(MRI)
* No distant metastasis
* Karnofsky score≥70
* Female patients need contraception during the test
* Postmenopausal women for at least 12 months, expect pregnancy possibility
* Patients did not receive chemotherapy, radiotherapy in any form before
* No other severe related diseases (such as other tumor, severe cardiac and central nervous system diseases, etc.)

Exclusion Criteria:

* Be treated by radiotherapy, chemotherapy or tumor biological therapy before
* Received immunosuppressive therapy (including corticosteroids)
* Participated in other clinical trial(s) in 1 month
* With malignant tumor of colon
* Peripheral neuropathy (WHO I level and above)
* Neurological or psychiatric abnormalities affecting cognition , including central nervous system metastasis
* Severe allergies or allergic history
* Severe pulmonary or heart disease
* Pregnant or lactation or refuse contraception during the test
* Suffering other malignant tumors in past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3-year

SECONDARY OUTCOMES:
Local recurrence rate | 3 years
Safety: Number of Participants with Adverse Events | 3 years
R0 resection rate | 1 year
Pathologic complete response | 1 year

OTHER OUTCOMES:
Compliance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Binbin Cui, MD, Principal Investigator — Department of Abdominal Surgery, Harbin Medical University Cancer Hospital
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China